CLINICAL TRIAL: NCT02836132
Title: Experience Success: Virtual Reality Skills Training to Enhance e-Weight Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Miriam Hospital (Other)
Collaborators: Virtually Better, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R42DK103537 (NIH)
Record Dates: First submitted 2016-07-14; First posted 2016-07-18 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Weight Watchers Online (Active Comparator): Participants will receive 6 months of no-cost access to the Weight Watchers Online platform.
  Interventions: Behavioral: Weight Watchers Online
- Weight Watchers Online + Experience Success (Experimental): Participants will receive 6 months of no-cost access to the Weight Watchers Online platform. They will also receive 6 months of no-cost access to the Experience Success online platform, with 4 virtual reality scenarios for training in behavioral weight loss skills.
  Interventions: Behavioral: Weight Watchers Online; Behavioral: Experience Success Virtual Reality Platform

INTERVENTIONS:
Behavioral: Weight Watchers Online
Behavioral: Experience Success Virtual Reality Platform
  Arms: Weight Watchers Online + Experience Success

SUMMARY:
The aim of this Phase II Small Business Technology Transfer grant is to complete development of a virtual reality intervention to augment and improve commercial Internet-delivered behavioral weight loss treatments, and to test it in a randomized controlled trial.

DETAILED DESCRIPTION:
Overweight and obesity are major health problems, affecting over two-thirds of US adults. Commercially available Internet-based weight loss programs are currently used by millions of overweight/obese individuals in the U.S, but weight losses are often poor, likely because these products on the whole do not incorporate empirically validated behavioral weight loss strategies that have been researched for over 40 years. Similarly, the weight losses obtained via research-based online weight loss programs are about half the size of those obtained via in-person treatment, likely because of the lack of (1) "hands-on" training in behavioral weight control strategies, and (2) support and guidance from group leaders and peers, both of which are hallmarks of traditional in-person treatment. The goal of this application is to improve commercial Internet -delivered behavioral obesity treatments by developing a virtual reality (VR) system that can be integrated into existing Internet weight control programs, such as Weight Watchers Online. The VR system will allow users to experience learning, implementing, and mastering behavioral weight control strategies in controlled virtual settings. The VR system will: (a) increase awareness of barriers to weight control behaviors, (b) teach skills to cope with these barriers, (c) build confidence using these skills, and (d) increase commitment to using these skills in real-world situations. The design of the VR System is based on Social Cognitive Theory, which states that health behaviors are learned by observing and imitating peers and role models, and by receiving social reinforcement. A randomized controlled trial (RCT) will be conducted with N = 125 participants to test the efficacy of 4 scenarios for improving weight losses obtained in a popular paid commercial weight loss program (Weight Watchers Online) over 6 months.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) 25-45 kg/m^2
* English speaking and literate
* able to walk 2 blocks unassisted without stopping
* access to a computer and the Internet

Exclusion Criteria:

* report of a heart condition, chest pain during periods of activity or rest, or loss of consciousness
* a medical condition that would affect the safety and/or efficacy of a weight management program involving diet and physical activity
* report of a condition that in the judgment of the Principal Investigator would render the participant potentially unlikely to be able to follow the study protocol for 6 months, including terminal illness, substance abuse, eating disorder, dementia, or other significant uncontrolled psychiatric problem
* currently pregnant, within 6-months postpartum, or intend to become pregnant within 6 months
* plan to move out of the local geographic area within 6 months
* previous participation in a weight loss study at the Weight Control and Diabetes Research Center of Brown University and The Miriam Hospital within the last 2 years
* current participation in another behavioral weight control program

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 3 months after beginning treatment
Weight loss | 6 months after beginning treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The Miriam Hospital Weight Control and Diabetes Research Center, Providence, Rhode Island, United States